CLINICAL TRIAL: NCT01414673
Title: Spontaneous Triggering of Ovulation vs. Administration of Human Chorionic Gonadotropin in Patients Undergoing Intrauterine Insemination: a Prospective Randomized Study.
Brief Title: HCG Versus Spontaneous LH in Intrauterine Insemination (IUI ) Cycles
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Devroey Paul, CRG
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: WAS11
Record Dates: First submitted 2011-08-05; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Spontaneous Triggering of Ovulation vs. Administration of Human Chorionic Gonadotropin in Patients Undergoing IUI
Keywords: IUI; HCG; Spontaneous LH; pregnancy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- spontaneous LH (Other)
  Interventions: Drug: HCG
- HCG (Experimental)
  Interventions: Drug: HCG

INTERVENTIONS:
Drug: HCG — 5000 IU

SUMMARY:
We recently reported the superiority of the natural cycle to a natural cycle controlled by the administration of human chorionic gonadotropin (hCG) for planning the frozen-thawed embryo transfer cycles, demonstrating a probable negative impact of exogenous hCG on endometrial receptivity.Based on the above findings we conducted the first prospective study that assesses whether there is a difference in pregnancy rate after intrauterine insemination (IUI) in a natural cycle with spontaneous luteinizing hormone (LH) rise compared to natural cycles controlled by hCG for final ovulation.

ELIGIBILITY:
Inclusion Criteria:

* age ≤ 36 years,
* regular menstrual cycles,
* body mass index (BMI) between 18 and 29 kg/m²,
* basal levels of FSH (≤ 12 IU/l),
* estradiol (≤ 80 pg/ml) and progesterone (≤ 1.6ng/ml) on day one of the cycle, normal hysterosalpingography (maximum 3 months prior starting the cycle).
* The use of donor sperm was also accepted as inclusion criteria.

Exclusion Criteria:

* PCOS
* endometriosis

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Uzbrussel, Brussels, Laarbeeklaan 101, Belgium

REFERENCES:
- [Result] Kosmas IP, Tatsioni A, Fatemi HM, Kolibianakis EM, Tournaye H, Devroey P. Human chorionic gonadotropin administration vs. luteinizing monitoring for intrauterine insemination timing, after administration of clomiphene citrate: a meta-analysis. Fertil Steril. 2007 Mar;87(3):607-12. doi: 10.1016/j.fertnstert.2006.10.003. Epub 2006 Dec 14. PMID 17173907
- [Derived] Kyrou D, Kolibianakis EM, Fatemi HM, Grimbizis GF, Theodoridis TD, Camus M, Tournaye H, Tarlatzis BC, Devroey P. Spontaneous triggering of ovulation versus HCG administration in patients undergoing IUI: a prospective randomized study. Reprod Biomed Online. 2012 Sep;25(3):278-83. doi: 10.1016/j.rbmo.2012.05.005. Epub 2012 May 23. PMID 22796236